CLINICAL TRIAL: NCT00877760
Title: Augmenting Response to Entecavir Using a Temporary Peginterferon Alpha-2a add-on Strategy for the Treatment of HBeAg-positive Chronic Hepatitis B
Brief Title: Augmenting Response to Entecavir With Peginterferon a-2a for the Treatment of HBeAg-positive Chronic Hepatitis B
Acronym: ARES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBV 09-01
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B Entecavir pegylated interferon a-2a
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ETV + pegIFN (Experimental): Patients receive Entecavir in a dosage of 0.5 mg once daily per os from day 0, up to week 48. From week 24 to week 48, they also receive pegylated-interferon a-2a in a dose of 180 μg per week s.c. At week 48, response will be assessed. Responders will continue to take Entecavir until week 72, and quit subsequently. Non-responders at week 48 will continue on Entecavir up to week 96.
  Interventions: Drug: pegylated interferon a-2a; Drug: Entecavir
- ETV (Active Comparator): Patients receive Entecavir in a dosage of 0.5 mg once daily per os from day 0, up to week 48. At week 48, response will be assessed. Responders will continue to take Entecavir until week 72, and quit subsequently. Non-responders at week 48 will continue on Entecavir up to week 96.
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: pegylated interferon a-2a — 180 μg, once per week s.c. for 24 weeks
  Other Names: Pegasys
  Arms: ETV + pegIFN
Drug: Entecavir — 0.5 mg once daily per os, either 72 weeks or 96 weeks
  Other Names: Baraclude

SUMMARY:
The purpose of this study is to investigate whether it is possible to augment the response of patients with HBeAg-positive chronic hepatitis B to entecavir by using a temporary peginterferon alpha-2a add-on strategy

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B (HBsAg positive > 6 months)
* HBeAg positive, anti-HBe negative at screening
* ALT > 1.3 x ULN within 60 days prior to screening and during screening
* Liver biopsy performed within 2 years prior to screening or during screening
* Age > 18 years
* Written informed consent
* Adequate contraception for males and females during treatment and follow up; negative pregnancy test (for women of childbearing potential)

Exclusion Criteria:

* Antiviral therapy against HBV within the previous 6 months
* Treatment with any investigational drug within 30 days of screening
* Previous treatment with lamivudine or telbivudine for more than six months
* Severe hepatitis activity as documented by ALT>10 x ULN
* History of decompensated cirrhosis (defined as jaundice in the presence of cirrhosis, ascites, bleeding gastric or esophageal varices or encephalopathy)
* Pre-existent neutropenia (neutrophils < 1,500/mm3) or thrombocytopenia (platelets < 90,000/mm3)
* Co-infection with hepatitis C virus or human immunodeficiency virus (HIV)
* Other acquired or inherited causes of liver disease (i.e. alcoholic liver disease, obesity induced liver disease, drug related liver disease, auto-immune hepatitis, hemochromatosis, Wilson's disease or alpha-1 antitrypsin deficiency)
* Alpha fetoprotein > 50 ng/ml
* Hyper- or hypothyroidism (subjects requiring medication to maintain TSH levels in the normal range are eligible if all other inclusion/exclusion criteria are met)
* Immune suppressive treatment within the previous 6 months
* Contra-indications for alpha-interferon therapy like suspected hypersensitivity to interferon or PEG-interferon or any known pre-existing medical condition that could interfere with the patient's participation in and completion of the study.
* Pregnancy, lactation
* Other significant medical illness that might interfere with this study: significant pulmonary dysfunction in the previous 6 months, malignancy other than skin basocellular carcinoma in previous 5 years, immunodeficiency syndromes (e.g. HIV positivity, auto-immune diseases, organ transplants other than cornea and hair transplant)
* Any medical condition requiring, or likely to require chronic systemic administration of steroids, during the course of the study
* Substance abuse, such as alcohol (> 80 g/day), I.V. drugs and inhaled drugs in the past 2 years.
* Any other condition which in the opinion of the principal investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in and completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2009-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The combined presence of HBV DNA level < 200 IU/mL and HBeAg loss | week 48

SECONDARY OUTCOMES:
ALT normalization | up to week 96
Undetectable HBV DNA <60 IU/mL | up to week 96
HBsAg and HBeAg loss from serum | up to week 96
The emergence of HBV polymerase mutations associated with reduced susceptibility to entecavir | up to week 96
Sustained response defined as the combined presence of HBV DNA level < 200 IU/mL and HBeAg loss | week 96

CONTACTS AND LOCATIONS:
Overall Officials: Harry Janssen, Prof. dr., Principal Investigator — Foundation for Liver Research (SLO) and Erasmus Medical Center
Locations (13):
- China (3):
  - Ruijin Hospital, Shanghai
  - Shanghai Public Health Center, Shanghai
  - Zhong Shan hospital, Fu Dan University, Shanghai
- Netherlands (2):
  - Amsterdam Medical Center (AMC), Amsterdam
  - Erasmus Medical Center, Rotterdam
- Poland (3):
  - CMUMU, Bydgoszcz
  - Medical University, Dept of Infections Diseases, Wroclaw
  - WAMED, Zawiercie
- Romania (2):
  - Fundeni Clinical Institute, Bucharest
  - Nat. Institute of inf. Disease, Bucharest
- Turkey (Türkiye) (3):
  - University of Ankara, Medical School, Ankara
  - Yuksek Ihsitas Hospital, Dept. Gastroenterology, Ankara
  - Cerrahpasa Medical Faculty, Istanbul

REFERENCES:
- [Derived] Brakenhoff SM, de Knegt RJ, van Campenhout MJH, van der Eijk AA, Brouwer WP, van Bommel F, Boonstra A, Hansen BE, Berg T, Janssen HLA, de Man RA, Sonneveld MJ. End-of-treatment HBsAg, HBcrAg and HBV RNA predict the risk of off-treatment ALT flares in chronic hepatitis B patients. J Microbiol Immunol Infect. 2023 Feb;56(1):31-39. doi: 10.1016/j.jmii.2022.06.002. Epub 2022 Jul 2. PMID 35941076
- [Derived] Brakenhoff SM, de Knegt RJ, Oliveira J, van der Eijk AA, van Vuuren AJ, Hansen BE, Janssen HLA, de Man RA, Boonstra A, Sonneveld MJ. Levels of Antibodies to Hepatitis B Core Antigen Are Associated With Liver Inflammation and Response to Peginterferon in Patients With Chronic Hepatitis B. J Infect Dis. 2022 Dec 28;227(1):113-122. doi: 10.1093/infdis/jiac210. PMID 35599306
- [Derived] Liem KS, van Campenhout MJH, Xie Q, Brouwer WP, Chi H, Qi X, Chen L, Tabak F, Hansen BE, Janssen HLA. Low hepatitis B surface antigen and HBV DNA levels predict response to the addition of pegylated interferon to entecavir in hepatitis B e antigen positive chronic hepatitis B. Aliment Pharmacol Ther. 2019 Feb;49(4):448-456. doi: 10.1111/apt.15098. PMID 30689258
- [Derived] Brouwer WP, Xie Q, Sonneveld MJ, Zhang N, Zhang Q, Tabak F, Streinu-Cercel A, Wang JY, Idilman R, Reesink HW, Diculescu M, Simon K, Voiculescu M, Akdogan M, Mazur W, Reijnders JG, Verhey E, Hansen BE, Janssen HL; ARES Study Group. Adding pegylated interferon to entecavir for hepatitis B e antigen-positive chronic hepatitis B: A multicenter randomized trial (ARES study). Hepatology. 2015 May;61(5):1512-22. doi: 10.1002/hep.27586. Epub 2015 Feb 27. PMID 25348661